CLINICAL TRIAL: NCT05799404
Title: Stapes Footplate Thickness Measured With UHR-CT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, GILLET Romain, MD, MSK Radiologist, Central Hospital, Nancy, France
Other Study IDs: N°3-RCB/EUDRACT
Record Dates: First submitted 2022-12-05; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Otosclerosis; Otitis Media
Keywords: ultra high resolution; ct; stapes; footplate; otosclerosis; otitis media
MeSH Terms: conditions — Otosclerosis; Otitis Media

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- otosclerosis: otosclerosis patients
  Interventions: Diagnostic Test: ultra-high resolution CT
- chronic otitis media: otitis media with middle ear opacities
  Interventions: Diagnostic Test: ultra-high resolution CT
- controls: sudden ear loss, pre-implantatory imaging, vertigo, tympanic perforation
  Interventions: Diagnostic Test: ultra-high resolution CT

INTERVENTIONS:
Diagnostic Test: ultra-high resolution CT — stapes footplate thickness measurement

SUMMARY:
The aim of this study is to compare the thickness of the stapes footplate measured with ultra high resolution CT in control patients, otosclerosis patients and chronic otitis media patients.

DETAILED DESCRIPTION:
Stapes footplate thickness will be measured under its anterior crus, its posterior crus and at its midpoint, in both the stapes axial plane and the laletral semi-circular canal planes.

ELIGIBILITY:
Inclusion Criteria:

* Ultra high resolution CT of the temporal bone available

Exclusion Criteria:

* previous surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients refered to our department between october 2020 and October 2022 for an ultra high resolution CT of the temporal bone
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-04-28 (Estimated); Primary Completion 2023-06-28 (Estimated); Study Completion 2023-06-28 (Estimated)

PRIMARY OUTCOMES:
stapes footplate thickness in mm in the stapes axial plane | october 2020-october 2022
  stapes footplate thickness measured with a digital caliper on our PACS system with the accuracy of a tenth of a millimetre, under the anterior crus of the stapes, under the posterior crus of the stapes, and at its midpoint, in the stapes axial plane and in the lateral semi circular canal plane, to compare both values and find out wich one is the most pertinent

SECONDARY OUTCOMES:
interobserver variability | october 2020-october 2022
  interobserver variability

CONTACTS AND LOCATIONS:
Overall Officials: romain gillet, MD, Principal Investigator — CHRU de Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akazawa Y, Ganaha A, Higa T, Kondo S, Oyakawa Y, Hirakawa H, Suzuki M, Yamashiro T. Measurement of stapes footplate thickness in otosclerosis by ultra-high-resolution computed tomography. Acta Otolaryngol. 2020 Nov;140(11):899-903. doi: 10.1080/00016489.2020.1788225. Epub 2020 Jul 23. PMID 32700991
- [Background] Tang R, Yin H, Wang Z, Zhang Z, Zhao L, Zhang P, Li J, Zhao P, Lv H, Zhang L, Yang Z, Wang Z. Stapes visualization by ultra-high resolution CT in cadaveric heads: A preliminary study. Eur J Radiol. 2021 Aug;141:109786. doi: 10.1016/j.ejrad.2021.109786. Epub 2021 May 21. PMID 34058698